CLINICAL TRIAL: NCT06851221
Title: Β3-adrenoreceptor As Prognostic Marker in Neuroblastoma and Ewing Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Maura Calvani, Head of Traslational oncoematology laboratory, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BETA3TumPed
Record Dates: First submitted 2025-02-21; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma; Ewing Sarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- biological samples analysis (Other)
  Interventions: Diagnostic Test: beta3 expression

INTERVENTIONS:
Diagnostic Test: beta3 expression — the samples leftover from the standard diagnostic procedures will be analyzed for the expression of the beta3-adrenoreceptor

SUMMARY:
This study on biological samples of patients affected by neuroblastoma and Ewing sarcoma aims at validating the beta3-adrenoreceptor as prognostic biomarker.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Ewing sarcoma or neuroblastoma

Exclusion Criteria:

* sieropositivity

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
expression of beta3-adrenoreceptor | from enrollment to the performance of the analysis that can take up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio traslazionale in oncoematologia, Florence, Italy, Italy